CLINICAL TRIAL: NCT03000296
Title: Autologous Unselected Hematopoietic Stem Cell Transplantation for Refractory Crohn's Disease
Acronym: AutoChron
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beneficência Portuguesa de São Paulo (Other)
Responsible Party: Principal Investigator, Milton Artur Ruiz, MD,PhD., Beneficência Portuguesa de São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: autocrohnproject1
Record Dates: First submitted 2016-12-09; First posted 2016-12-22 (Estimated); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Crohn's Disease; Inflammatory Bowel Diseases; Gastroenteritis
Keywords: autologous; lymphoablation; hematopoetic stem cell transplant; immune system; Bone marrow transplant
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases; Gastroenteritis | interventions — Bone Marrow Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hematopoietic Stem Cell Transplantation (Experimental): High doses immunosuppression Cyclophosphamide (200 mg/kg total dose for four days) and rabbit antithymocyte globulin (6.5 mg/kg total dose for four days) followed by unselected autologous hematopoietic stem cell transplantation rescue.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Hematopoietic stem cell transplantation Lymphoablation followed by hematopoietic stem cell transplantation to rescue the immune system.
  Other Names: Bone Marrow Transplantation; Hematopoietic Stem Cell Transplatation

SUMMARY:
This study evaluates the safety and clinical benefits of a therapeutic approach using the cyclophosphamide (Cy) + thymoglobulin® (ATG) + granulocyte colony-stimulating factor (G-CSF) conditioning regimen followed by autologous hematopoietic stem cell transplantation (HSCT) rescue in the treatment of refractory Crohn's disease. Adverse events, and clinical and endoscopic conditions will be assessed at different short and long-term time points.

DETAILED DESCRIPTION:
Crohn's disease (CD) is a chronic, refractory inflammatory bowel disease that affects the entire digestive tract associated with intestinal and extra intestinal manifestations or other autoimmune diseases. Conventional therapy for Crohn's disease includes anti-inflammatory, immunosuppressant and/or biologic drugs/corticosteroids. This treatment benefits the majority of patients. However, a proportion of patients fail to achieve complete and long-term disease control and often require multiple intestinal surgeries with a risk of developing short bowel syndrome.

Hematopoietic stem cell transplantation (HSCT) has been proposed to cause lymphoablation and reset of the immune system as an alternative strategy to induce long-term disease control in this high-risk population.

This study enrolled Crohn's disease patients not responsive to conventional therapy.

Initially safety and the clinical outcome will be evaluated. The selected patients will be admitted to the bone marrow transplant (BMT) unit for the mobilization regimen using cyclophosphamide (Cy - 60 mg/kg) and G-CSF (10 mcg/kg/day) from the 5th day after Cy administration until harvesting progenitor cells from peripheral blood by leukapheresis.

After seven days of rest, the conditioning regimen consists of Cy (200 mg/kg total dose for four days), rabbit antithymocyte globulin (6.5 mg/kg total dose for four days) and methylprednisolone (500 mg/day).

The clinical course of patients with refractory Crohn´s disease will be evaluated to determine the efficacy of HSCT as a therapeutic tool including the adverse aspects of the procedure, clinical outcome and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 14 and 50 years (patients aged 50 - 70 can participate at the principal investigators discretion).
2. Confirmed diagnosis of active Crohn's disease:

   * Diagnosis of Crohn's disease based on typical radiological findingsand or typical histology at least 6 months prior to screening.
   * Active disease at the time of registration to the trial, defined as

     *Crohn's Disease Activity Index (CDAI) > 150, and ii) Two of the following:
   * Harvey Bradshaw Index > 4
   * Endoscopic evidence of active disease confirmed by histology
   * Clear evidence of active small bowel Crohn's disease on computed tomography (CT) or magnetic resonance (MR) enterography.
3. Unsatisfactory course despite immunosuppressive agents (usually azathioprine, methotrexate and two biologic agents (normally infliximab, adalimumab and/or certolizumab) in addition to corticosteroids. Patients should have relapsing and refractory disease despite thiopurines, methotrexate and/or infliximab/adalimumab/certolizumab maintenance therapy or clear demonstration of intolerance / toxicity to these drugs.
4. Current problems unsuitable for surgery or patient at risk for developing short bowel syndrome.
5. Informed consent:

   * Prepared to undergo additional study procedures as per trial schedule
   * Patient has undergone intensive counseling about risks

Exclusion Criteria:

1. Pregnancy or unwillingness to use adequate contraception during the study, in women of childbearing age. Unwillingness of using appropriate contraceptive measures in males.
2. Concomitant severe disease

   * renal: creatinine clearance < 30 mL/min (measured or estimated)
   * cardiac: clinical evidence of refractory congestive heart failure; left ventricular ejection fraction < 40% by multigated radionuclide angiography (MUGA) or cardiac echo; chronic atrial fibrillation necessitating oral anticoagulation; uncontrolled ventricular arrhythmia; pericardial effusion with hemodynamic consequences as evaluated by an experienced echo cardiographer.
   * pulmonary: diffusion capacity <40%
   * psychiatric disorders including active drug or alcohol abuse
   * concurrent or recent history of malignant disease (excluding non-melanoma skin cancer)
   * uncontrolled hypertension, defined as resting systolic blood pressure ≥ 140 and/or resting diastolic pressure ≥ 90 despite at least 2 anti-hypertensive agents.
   * uncontrolled acute or chronic infection with HIV, Human T-lymphotropic virus (HTLV-1 or 2), hepatitis viruses or any other infection the investigators consider a contraindication to participation.
   * other chronic disease causing significant organ failure.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-10; Primary Completion 2017-12 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Safety of unselected autologous HSCT in refractory Crohn´s disease patients | 12 months
  HHSCT safety will be analyzed by laboratory tests and treatment-related adverse events. Safety will be evaluated by treatment-related adverse events. All adverse events will be recorded in a standardized way and their relationship to the study protocol will be assessed at different short- and long-term time points.

SECONDARY OUTCOMES:
Crohn´s Disease Activity Index (CDAI) | 12 months
  Duration of disease remission, defined as a CDAI ≤ 150, will be assessed at 1, 3, 6, 12 and 24 months after transplant.
CRAIG Crohn´s Severity Score (CSS) | 12 months
  The CRAIG CSS will be assessed at 1, 3, 6, 12 and 24 months after transplant.
Inflammatory Bowel Disease Questionnaire (IBDQ) | 24 months
  The IBDQ will be administered at 1, 3, 6, 12 and 24 months after transplant.
Short Form-36 Health Survey (SF-36) | 24 months
  The SF-36 will be administered at 1, 3, 6, 12 and 24 months after transplant.
Simple Endoscopic Activity Score (SES) | 24 months
  The SES will be assessed at 6, 12 and 24 months after HSCT.
Crohn's Disease Endoscopic Index of Severity (CDEIS) | 24 months
  The CDEIS will be assessed at 6, 12 and 24 months after HSCT.
Rutgeerts endoscopic score | 24 months
  Rutgeerts endoscopic score will be assessed at 6, 12 and 24 months after HSCT.
Harvey & Bradshaw Index (HBI) | 24 months
  The HBI will be assessed at 1, 3, 6, 12 and 24 months after HSCT.

CONTACTS AND LOCATIONS:
Overall Officials: Milton A Ruiz, MD, PhD, Principal Investigator — Beneficencia Portuguesa
Locations (1):
- Beneficencia Portuguesa, São José do Rio Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The main objective is to observe the safety and clinical benefit of autologous HSCT therapy in refractory patients with Crohn's disease. Evaluation during transplant period and 1, 3, 6, 12 and 24 months post-transplant. Safety be evaluated by the amount of treatment-related adverse events. Record adverse events in a standardized way. Secondary outcome measures will be disease remission: 1, 3, 6, 12 and 24 months post-transplant both clinical and endoscopic remission. The percentage of patients in sustained disease remission at 1, 3, 6, 12 and 24 months post HSCT will be determined. Sustained disease remission is defined as a CDAI < 150; HBI <4, CCSI< 16, without the use of corticosteroids, immunosuppressant or biologic agents. Mucosal healing will be assessed during ileocolonoscopy at 6, 12, and 24 months following HSCT using SES, CDEIS and Rutgeerts endoscopy index. Heath Quality life, Short Form 36 and IBDQ at 1 3 6 12 and 24 months post-Transplant.